CLINICAL TRIAL: NCT05959785
Title: Diaphragmatic Exercises As Treatment of Referred Pain After Total Laparoscopic Hysterectomy: Randomized Controlled Clinical Trial.
Brief Title: Diaphragmatic Exercises As Treatment of Referred Pain After Total Laparoscopic Hysterectomy: Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Antonio Luis Partida Márquez, Diplomado en Enfermería, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALPM21
Record Dates: First submitted 2023-03-30; First posted 2023-07-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hysterectomy
Keywords: pain; phrenic nerve; shoulder; laparoscopy
MeSH Terms: conditions — Pain | interventions — Alkalies; Control Groups

STUDY DESIGN:
Intervention Model Description: Clinical trial with control group and random assignment intervention
Who Masked: Participant
Masking Description: plain blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Assignment to the intervention group will be done by simple randomization of the sample. A random sequence of numbers will be generated using the statistical program SPSS v.28. Patients will be included in the intervention group of each subcategory if their subject number matches one of the random numbers generated.The intervention groups will receive an explanatory video where a study collaborator performs a series of abdominal or diaphragmatic breathing exercises, which are intended to assess their effectiveness in this clinical trial.
  Interventions: Procedure: Abdominal or diaphragmatic breathing exercises
- control groups (Placebo Comparator): The patients belonging to the control groups of each subcategory will also receive an explanatory video with basic and light cervical mobilization exercises (Annex 12). This group of exercises will be made up of a series of cervical mobilization exercises that are performed without pain, smooth, controlled by the patients, and without forcing the angulations. They are performed seated, with the arms extended along the body and forearms and hands resting on the legs. The chair must be firm and comfortable. Head movements to the right and left, right and left lateral flexion of the cervical region, cervical flexion and extension will be performed. This exercise will be performed for 5 minutes 3 times a day and beginning in the first 24 postoperative hours.
  Interventions: Procedure: Basic and light cervical mobilization exercises

INTERVENTIONS:
Procedure: Basic and light cervical mobilization exercises — This group of exercises will be made up of a series of cervical mobilization exercises that are performed without pain, smooth, controlled by the patients, and without forcing the angulations. They are performed seated, with the arms extended along the body and forearms and hands resting on the legs. The chair must be firm and comfortable. Head movements to the right and left, right and left lateral flexion of the cervical region, cervical flexion and extension will be performed. This exercise will be performed for 5 minutes 3 times a day and beginning in the first 24 postoperative hours.
  Other Names: Control group
  Arms: control groups
Procedure: Abdominal or diaphragmatic breathing exercises — The first abdominal or diaphragmatic breathing exercises will be carried out in a lying position, with the back well supported on a comfortable and firm surface, and with hips and knees flexed and feet supported. The patients take deep breaths, taking air raising the abdomen towards the ceiling, without raising the back from the horizontal plane. During expiration the navel will lower posteriorly and rise towards the thoracic region. For the second abdominal or diaphragmatic breathing exercise, the patient is seated on a firm and comfortable surface, with hips and knees flexed and feet supported. An inspiratory movement will be made in which the patient's navel will be moved outward, away from the spine. During expiration, the navel will go in the direction of the patient's spine and will rise in the direction of the thorax.
  Other Names: Intervention group
  Arms: intervention group

SUMMARY:
Through a blinded clinical trial, the aim is to evaluate the efficacy of manual therapy in the treatment of pain referred to after laparoscopic hysterectomy.

Control and intervention groups were randomly established. Informed consent will be requested for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who have given their consent to participate in the project by signing the informed consent.

  * Patient between 18 and 65 years of age.
  * Patients with a hysterectomy scheduled to be performed in less than 3 months at the Women's Hospital in Seville or at the Quirón Sagrado Corazón Clinic in Seville.
  * Who develops pain of intensity greater than 7 points located in the head, neck or upper limbs in the first 24 hours post-hysterectomy.
  * Patients who are able to communicate in Spanish or English.

Exclusion Criteria:

* Neurological Pathology.
* Non-cooperative Subject.
* Severe Psychiatric Illness.
* Loss of Cognitive Capacity.
* Evidence that post-hysterectomy pain is not caused by surgery (eg, presence of fracture or infection in the head, neck or upper limbs.
* Localized pain in areas not considered in this study and that may affect the performance and results of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
The McGill Pain Questionnaire | 24 hours after laparoscopy
  Location of pain: which is usually represented by a schematic figure of the human body, where the patient points out the areas where they feel pain.
  * Quality of pain: the patient must choose from a wide list of types of pain those characteristics that define the one he presents. They are grouped into various categories that in turn form four large groups: sensory, emotional, evaluative and miscellaneous. In the original English version, the number of words was 78, although they may vary in the different validations of the questionnaire (66 in the Spanish version).
  * Pain intensity at the current moment: explored by means of a question with five possible response categories.
  * Assessment of pain at the current time using a visual analogue scale, ranging from "no pain" to "unbearable pain".
The Brief Pain Questionnaire | 24 hours after laparoscopy
  This questionnaire, in its short version, includes a body map that the patient can use to mark the areas where pain is located. In addition to providing a useful tool for localizing pain, this questionnaire provides important information about other characteristics of pain, as well as response to prescribed treatments.
The Quick Dash quiz | 24 hours after laparoscopy
  Questionnaire containing questions about symptoms and the ability to use instruments of the upper limbs. Collect data referring to the last week
The HIT-6 scale | 24 hours after laparoscopy
  evaluates the headache through 6 questions
The Neck Disability Index questionnaire | 24 hours after laparoscopy
  assesses neck and back pain and its influence on basic activities of daily living

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Quiron Sagrado Corazon, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No